CLINICAL TRIAL: NCT04258774
Title: The Effect of Respiratory Challenge on the BOLD Signal
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201910105
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypoxia, Brain; Hyperoxia; Hypercapnia; Hypocapnia
Keywords: brain metabolism; oxygen extraction fraction; cerebral vascular reactivity; carbon dioxide
MeSH Terms: conditions — Hypoxia, Brain; Hyperoxia; Hypercapnia; Hypocapnia | interventions — Carbon Dioxide

STUDY DESIGN:
Intervention Model Description: All arms will receive the same study conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Adults (Active Comparator)
  Interventions: Other: Carbon Dioxide
- Adults diagnosed with vascular pathology of the brain (Active Comparator)
  Interventions: Other: Carbon Dioxide

INTERVENTIONS:
Other: Carbon Dioxide — The study team will administer inhaled carbon dioxide to the participants during an MRI at a level

SUMMARY:
The purpose of this research study is to better understand how blood flow and metabolism are different between normal controls and patients with disease.

The investigators will examine brain blood flow and metabolism using magnetic resonance imaging (MRI). The brain's blood vessels expand and constrict to regulate blood flow based on the brain's needs. The amount of expanding and contracting the blood vessels can do varies by age. The brain's blood flow changes in small ways during everyday activities, such as normal brain growth, exercise, or deep concentration. Significant illness or physiologic stress may increase the brain's metabolic demand or cause other bigger changes in blood flow. If blood vessels are not able to expand to give more blood flow when metabolic demand is high, the brain may not get all of the oxygen it needs. In less extreme circumstances, not having as much oxygen as it wants may cause the brain to grow and develop more slowly than it should.

One way to test the ability of the blood vessels to expand is by measuring blood flow while breathing in carbon dioxide (CO2). CO2 causes blood vessels in the brain to dilate without increasing brain metabolism. The study team will use a special mask to control the amount of oxygen and carbon dioxide patients breath in so that we can study how their brain reacts to these changes. This device designed to simulate carbon dioxide levels achieved by a breath-hold and target the concentration of carbon dioxide in the blood in breathing patients. The device captures exhaled gas and provides an admixture of fresh gas and neutral/expired gas to target different carbon dioxide levels while maintaining a fixed oxygen level. The study team will obtain MRI images of the brain while the subjects are breathing air controlled by the device.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects (>18 years old) OR adult patients (>18 years old) diagnosed with vascular pathology of the brain willing to participate and sign a consent form.
2. Able to participate in MRI scan without sedation
3. Not on stimulant medications
4. No psychiatric history, as defined by seeing a psychiatrist for medical evaluation and treatment, or taking anti-depressant medications
5. No seizure history
6. May have occasional headaches if not taking a daily preventative medication for headaches
7. Not on vasodilatory medication, such as sildenafil or verapamil

Exclusion Criteria:

1. Subjects refusing to undergo testing
2. Subjects with obstructive or resistive lung disease whose PaCO2 at rest is greater than 50mmHg or whose venous serum bicarbonate is greater than 26 mEq/L
3. Subjects with pre-existing respiratory or metabolic acidosis
4. Subjects who require portable oxygen at rest or with exercise
5. Subjects with chronic heart failure or severe pulmonary disease who are unable to climb one flight of stairs due to shortness of breath
6. Subjects with severe heart failure or restrictive lung disease with resting respiratory rate over 15 breaths/min 2. Patients that cannot participate in a course of rehabilitation therapy.
7. Subjects that cannot undergo an MRI scan due to one of the following indications:

   * Pregnancy
   * Obtundation, or Coma
   * Confusion, Delirium, or Dementia
   * Unable to understand or carry out commands regarding keeping still and breathing pattern
   * Increased intracranial pressure due to space occupying lesion or obstruction of outflow of CSF
   * Claustrophobia
   * History of kidney problems
   * Pace makers
   * Skin tattoos
   * Neurostimulators (TENS-unit)
   * Implanted drug infusion device (i.e., insulin pump)
   * Exposure of metal fragments to your eye
   * Artificial heart valves
   * Aneurysm clips
   * Cochlear implants
   * Metallic implants and prosthesis
   * Vascular stent or stent graft
   * History as a metal worker
   * Shrapnel or bullet wounds
   * Dorsal column stimulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral Oxygen Metabolism | From the beginning of the MRI scan to the completion of the MRI scan -- 75 minutes.

SECONDARY OUTCOMES:
Cerebrovascular Reactivity | From administration of carbon dioxide to end of inhalation of carbon dioxide -- 15 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University of St. Louis, St Louis, Missouri, United States